CLINICAL TRIAL: NCT07169110
Title: Study of the Interprofessional Reproducibility of a Clinical Observation Scale for the Development of Very Premature Infants Aged 1 to 6 Months Corrected, for the Very Early Detection of Developmental Disorders.
Brief Title: Study of the Interprofessional Reproducibility of a Clinical Observation Scale for the Development of Very Premature Infants
Acronym: SPIN-NA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0578; ID-RCB : 2025-A00379-40 (Other: ANSM)
Record Dates: First submitted 2025-08-01; First posted 2025-09-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prematurity
Keywords: Premature infant; early development; early care intervention; early evaluation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPIN-NA Evaluation: Infants evaluated by SPIN-NA grid
  Interventions: Other: SPIN-NA Developmental Observation Grid Assessment via Home-Based Standardized Video Recording

INTERVENTIONS:
Other: SPIN-NA Developmental Observation Grid Assessment via Home-Based Standardized Video Recording — The SPIN-NA intervention consists of an analytical assessment of development using a standardized clinical observation grid.
  Infants are filmed at home once between 1 and 6 months of corrected age in their family environment by the creators of the grid.
  The filmed observation includes structured observation scenarios designed to assess eight areas of development:
  stress signals, physiological and tonic regulation, perceptual abilities of different sensory channels, exploratory appetite, manipulative activities, child interactions and communication, emotional expressions and expressiveness, parent-child interactions: parental adaptation to the child's behavior.The videos are evaluated independently by five experienced psychomotor therapists trained together in the use of the SPINNA grid. No treatment or physical intervention is administered; the intervention is observational and non-invasive, aimed at validating the reproducibility of the grid in a real-world context.

SUMMARY:
The research concerns the study of the interprofessional reproducibility of a grid for observing the development of premature infants from 1 to 6 months corrected age. No tool is available to characterize the mechanisms of early developmental processes and their deviations. We propose an analytical observation grid of developmental mechanisms in the first few months, in order to identify warning signs of developmental deviations and help define the nature and type of early care for vulnerable infants.

DETAILED DESCRIPTION:
Improving the development of premature babies is a challenge. Developmental disabilities are common. Brain damage accounts for only a small proportion of disorders. Other factors have a major influence on the outcome: immaturity, an intrusive and stressful hospital environment, and parental socio-psychological conditions. Early sensory-motor disorders disrupt development. The high degree of cerebral plasticity in infants means that early care is essential if developmental trajectories are to be improved. Intervention programmes are heterogeneous. Meta-analyses therefore make only limited comparisons. The cognitive and behavioural benefits are variable. Motor benefits are low. No tools are available to determine the mechanisms of early developmental processes.

The SPIN-NA grid is a scale for analytical observation of developmental processes from 1 to 6 months corrected age to identify early warning signs and determine early care (nature, areas of care, objectives). The aim is to study the inter-professional reproducibility of the grid. This validation stage is essential if the grid is to serve as a reference tool in psychomotricity for vulnerable newborns.

Premature babies born between 27 and 32 gestational weeks will be assessed using the SPIN-NA grid by 5 experienced psychomotor-therapists, on the basis of videos taken at home between 1 and 6 months corrected age, by the creators of the grid. Each child was filmed only once. The inter-observer agreement should be at least 70% for the 8 observation axes defined in the SPIN-NA grid.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child born between 27 and 32 weeks of amenorrhea in a singleton pregnancy;
* Child hospitalized in the neonatology unit of Toulouse University Hospital;
* Family home within a 15 km radius of Toulouse to allow for home visits for filming;
* Parents with parental authority affiliated with a social security scheme or equivalent;
* Signature of the informed consent form by the parents with parental authority
* Absence of serious illness, as defined in the exclusion criteria;
* The child may participate in another study during the duration of this study, without an exclusion period.

Exclusion Criteria:

* Child with a severe organic pathology detected during hospitalization and requiring specific and appropriate care for the diagnosed pathology;
* Child with a neurological complication: Grade 3 or 4 intraventricular hemorrhage, periventricular cavitary leukomalacia, excluding frontal leukomalacia;
* Child with a malformation or multiple malformations that impair the neurological prognosis;
* Child with genetic or metabolic diseases;
* Fetal alcohol syndrome;
* Parental authority holders under guardianship, curatorship, or legal protection;
* Any family condition that prevents compliance with the procedures set out in the study protocol, in the opinion of the investigator.
* Family members who do not speak French fluently, in order to ensure understanding of the system and the proposed care.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be selected from infants born and hospitalized in the neonatology department of Toulouse University Hospital. The study targets a local population, with families residing within a 15-kilometer radius of Toulouse to allow for home-based video recording.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Inter-Rater Agreement on Developmental Difficulties Detection Using the SPIN-NA Grid Across 8 Observation Axes | At the day 1 corresponding to the home video recording
  The primary outcome is the overall percentage of agreement between raters, calculated as the mean of agreement rates across all evaluator pairs. Agreement is defined as both raters assigning the same classification (presence or absence of anomaly) to a given infant for a given axis.

SECONDARY OUTCOMES:
Inter-Rater Agreement on SPIN-NA Grid Evaluations by Age Group at the time of evaluation : 1-3 Months vs. 4-6 Months Corrected Age | At the day 1 corresponding to the home video recording
  Inter-rater agreement will be assessed separately for two age groups of infants: 1-3 months and 4-6 months corrected age. Each of the five trained psychomotor therapists will independently evaluate all infants in both age groups using the SPIN-NA grid. For each developmental axis, agreement is defined as two raters assigning the same classification (presence or absence of anomaly) to the same child. Agreement will be expressed as the mean percentage of agreement across all evaluator pairs for each age group. This analysis aims to explore whether the reproducibility of SPIN-NA assessments varies depending on the infant's age at the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Corine Alberge, Study Director — University Hospital of Toulouse; Nathalie Noack, Study Director — University Hospital of Toulouse
Locations (1):
- Intensive care /neonatology Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No